CLINICAL TRIAL: NCT02310698
Title: Comparison of Whole Breast Screening Ultrasound and Contrast Enhanced Mammography for Supplemental Breast Cancer Screening
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-240
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Screening
Keywords: Ultrasound; Enhanced Mammography; 14-240

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Breast Cancer Screening Patients: * Women presenting for screening full field digital mammography (FFDM) and WBUS on the same day or within 30 days of one another.
    o These women will be offered CEDM instead of the FFDM.
  * Women that are scheduled for CEDM alone.
    o These women will be offered WBUS in addition to the CEDM.
  * Women scheduled for both CEDM and WBUS on the same day or within 30 days of one another.
  Interventions: Device: contrast enhanced digital mammography (CEDM); Device: whole breast screening ultrasound (WBUS)

INTERVENTIONS:
Device: contrast enhanced digital mammography (CEDM)
Device: whole breast screening ultrasound (WBUS)

SUMMARY:
Breast tumors are often detected on mammography but may be harder to see in women with dense breasts. This is why screening breast ultrasound is sometimes used as another test in women with dense breasts. Ultrasound has been shown to detect additional cancers that are not seen on regular mammography.

Contrast Enhanced Digital Mammography (CEDM) is a FDA approved form of mammography. It is essentially a routine digital mammogram performed after iodine dye (the same that is used with CT scans) is injected into a vein in the arm. Like screening ultrasound, CEDM has been shown to detect breast cancers that are not seen on a regular mammogram. The purpose of this study is to compare whether CEDM or screening breast ultrasound is better at detecting cancer. Both will be done in this study and compared to one another.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for screening WBUS and a screening FFDM on the same day or within the following 30 days of each other
* Women scheduled for screening CEDM alone
* Women scheduled for WBUS and screening CEDM on the same day or within 30 days of one another

Exclusion Criteria:

* Age < 30 years old
* Male patients
* Patients with any clinical breast symptoms (palpable mass, nipple discharge, etc)
* Patients with known diagnosis of breast cancer
* Patients with any breast surgery or biopsy within 90 days prior to the study
* Patients who have had a lumpectomy for breast cancer within 18 months prior to the study
* Patients who are thought to have a breast MRI within 1 year prior to the study
* Patients with contraindication to the intravenous use of iodinated contrast agent (i.e. allergy to iodinated contrast or severely impaired renal function with a creatinine level ≥1.3)

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinic
Sampling Method: Non-Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2014-12-02 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
The number of cancers and false positive findings identified on a CEDM and WBUS as a measure of sensitivity and specificity. | 1 year
  With respect to imaging, a positive test is defined by a recommendation for biopsy (BIRADS 4 or 5). Negative imaging tests are those with BIRADS 1-3. The number of recommendations for short term follow up (BI-RADS 3) will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Sung, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Horvat JV, Amir T, Watt GP, Comstock CE, Nissan N, Jochelson MS, Sung JS. Comparison of Contrast-enhanced Mammography and Low-Energy Imaging with or without Supplemental Whole-Breast US in Breast Cancer Detection. Radiology. 2025 Mar;314(3):e242006. doi: 10.1148/radiol.242006. PMID 40067106
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/